CLINICAL TRIAL: NCT04670003
Title: Spread Analysis of COVID-19 Outbreak in France by Self-assessment Web-application: an Observational Study
Brief Title: Spread Analysis of COVID-19 Outbreak in France by Self-assessment Web-application
Acronym: SourceCOVID
Status: Completed | Type: Observational
Sponsor: Weprom (Other)
Collaborators: Kelindi (Industry)
Responsible Party: Sponsor
Other Study IDs: WP-2020-05
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- users: users of web-application
  Interventions: Other: users

INTERVENTIONS:
Other: users — Data of users of the web-application

SUMMARY:
A coronavirus pandemic began on 12/31/2019 with a first Chinese patient. As of 04/04/2020, the epidemic affects more than 190 countries with more than 50 million official contaminations and 1,251,000 deaths. (Univ J Hopkins). This virus causes a pathology ranging from simple flu-like symptoms in 80% of cases to acute respiratory distress syndromes requiring intensive care in 5% of cases and a death rate of 1.4 to 4% of cases.

Viral contamination is airborne and fecal A first epidemic wave crossed France in March / April 2020 then a second in October / November with a source of contamination which began in mid-August 2020. The sources of propagation are not well known (what places, what times, what contacts…? ) In the context of the health crisis linked to the coronavirus, knowledge of the sources of propagation of this 2nd wave is an important issue to guide end of lockdown and second lockdown policies.

ELIGIBILITY:
Inclusion criteria:

* users of the application
* not having objected to the use of their data

Exclusion criteria:

- user who does not have a complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All users of the application contaminated with COVID 19 who have not objected to the use of their data
Sampling Method: Non-Probability Sample
Enrollment: 4975 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Description of the methods of contamination of patients | 2 months
  Data and symptomes collected by the web applications self-questionnaire (patient reported outcome)

SECONDARY OUTCOMES:
Evaluation in time of the spread of the virus during the 2nd epidemic wave. | 2 months
  Data and symptomes collected by the web applications self-questionnaire (patient reported outcome)
Evaluation in space of the spread of the virus during the 2nd epidemic wave. | 2 months
  Data and symptomes collected by the web applications self-questionnaire according to ZIP code (patient reported outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DENIS, MD, Study Director — Institut Interrégional de Cancerologie et Kelindi
Locations (1):
- Institut Interrégional de Cancérologie, Le Mans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denis F, Septans AL, Le Goff F, Jeanneau S, Lescure FX. Analysis of COVID-19 Transmission Sources in France by Self-Assessment Before and After the Partial Lockdown: Observational Study. J Med Internet Res. 2021 May 4;23(5):e26932. doi: 10.2196/26932. PMID 33878018